CLINICAL TRIAL: NCT03193450
Title: Telephone-Based Re-Education of Drug Administration for Helicobacter Pylori Eradication: a Multi-Center Randomized, Controlled Study
Brief Title: Telephone-Based Re-education for Hp Eradication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, He Shuixiang, Director of the Department of Gastroenterology, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: XAJTU-DG001
Record Dates: First submitted 2017-06-17; First posted 2017-06-20 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: helicobactor pylori

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Re-education group (Experimental): Patients in this arm will receive a repeated instruction by telephone in terms of both calling and message at the forth, seventh, tenth day after the start of treatment.
  Interventions: Behavioral: telephone-based re-education; Behavioral: First education at the clinic
- Non re-education group (Active Comparator): Patients in this arm only received an instruction card about the drug administration at the clinic by doctors but no re-education by telephone during treatment
  Interventions: Behavioral: First education at the clinic

INTERVENTIONS:
Behavioral: telephone-based re-education — Patients will receive a repeated instruction by telephone in terms of both calling and message at the forth, seventh, tenth day after the start of treatment.
  Arms: Re-education group
Behavioral: First education at the clinic — Patients will receive an instruction card about the drug administration at the clinic by doctors.

SUMMARY:
It was suggested that the patient compliance plans an important role in the Hp eradication. However, data on whether re-education could improve the eradication rate are lacking. We consider that re-education on patients by telephone during the process of drug administration could increase the eradication rate in Hp infected patients.

We hypothesized that telephone re-education during the whole process of drug administration would improve the compliance of patients and ultimately increase the Hp eradication rate.

ELIGIBILITY:
Inclusion Criteria:

1. Prior informed consent
2. 18-70 years of age
3. Hp infected patients diagnosed by 13C urea breath test, including digestive ulcer, gastritis with dyspepsia symptoms, family history of gastric cancer, planning to use long-term non-steroidal anti-inflammatory drugs (NSAIDs), or personal request
4. Ability to swallow oral medications
5. No contraindication for the drugs used for Hp eradication
6. Both men and women enrolled in this trial must use adequate barrier birth control during the course of the trial and 4 weeks after the completion of trial

Exclusion Criteria:

1. Pregnant or breast-feeding subjects
2. Previous failed treatment of Hp eradication
3. Previous treatment with bismuth salts or antibiotics within 1 month before study enrollment, and treatment with proton pump inhibitor or H2 receptor antagonist within 2 weeks before study enrollment
4. Any disease that could jeopardize the safety of subject and their compliance in the study (e.g. serious liver disease, heart disease, kidney disease, malignant tumor or alcoholism, etc.)
5. Previous upper gastrointestinal surgery
6. Inability to express complaint (e.g. mental disorder, psychoneurosis, unable to cooperation, etc.)
7. Active clinically serious infections, except for Hepatitis B virus and hepatitis C virus infection
8. Clinically significant gastrointestinal bleeding within 4 weeks prior to start of study drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Hp eradication rate | 4-6 weeks after the end of drug administration
  Eradication rate is the proportion of patients with eradicated-Hp. Hp infection was considered eradicated when negative results were obtained by 13carbon urea breath test at 4-6 weeks after the end of drug administration

SECONDARY OUTCOMES:
Symptoms relief rate | 4-6 weeks after the end of drug administration
  The symptoms were recorded according to Gastrointestinal Symptom Rating Scale.
Adverse events | 4-6 weeks after the end of drug administration
  The terms and grade of adverse events will be presented according to the Common Terminology Criteria for Adverse Events (CTCAE: version 4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Shuixiang He, MD, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McColl KE. Clinical practice. Helicobacter pylori infection. N Engl J Med. 2010 Apr 29;362(17):1597-604. doi: 10.1056/NEJMcp1001110. No abstract available. PMID 20427808
- [Background] Malfertheiner P, Sipponen P, Naumann M, Moayyedi P, Megraud F, Xiao SD, Sugano K, Nyren O; Lejondal H. pylori-Gastric Cancer Task Force. Helicobacter pylori eradication has the potential to prevent gastric cancer: a state-of-the-art critique. Am J Gastroenterol. 2005 Sep;100(9):2100-15. doi: 10.1111/j.1572-0241.2005.41688.x. PMID 16128957
- [Background] Svedlund J, Sjodin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. 1988 Feb;33(2):129-34. doi: 10.1007/BF01535722. PMID 3123181